CLINICAL TRIAL: NCT01058603
Title: Multicentre, Randomised, Controlled Clinical Study on the Efficacy in Terms of Clinical Pregnancy Rate of 1 Embryo Transfer at Day 5 After Co-culture on Autologous Endometrial Cells(ENDOCELL®) Versus 1 Embryo Transfer at Day 3 After Culture on Conventional Medium.
Brief Title: Efficacy of Endocell® vs Conventional Medium in the Treatment of Infertility
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratoires Genévrier (Industry)
Responsible Party: Laboratoires Genévrier
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07F/END01
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Infertility
Keywords: Infertility; Cell Culture; AECC; Endocell; IVF
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- D3 (Active Comparator)
  Interventions: Other: - Conventional culture medium for IVF
- D5 (Experimental)
  Interventions: Other: - Endocell®

INTERVENTIONS:
Other: - Conventional culture medium for IVF — Embryos are cultured on conventional medium and transferred at Day 3. Supernumerary good quality embryos are frozen
  Arms: D3
Other: - Endocell® — Embryos are cultured on ENDOCELL® from Day 2 to Day 5 (Blastocyst stage) One embryo is transferred at Day 5. Supernumerary good quality embryos are frozen.
  Arms: D5

SUMMARY:
The aim of this study is to demonstrate the efficacy of a single embryo transfer at blastocyst stage (Day 5) after co-culture on Autologous Endometrial Cell Culture (AECC) versus transfer of a single embryo at Day 3 after culture in conventional medium. Efficacy will be assessed in terms of clinical pregnancy rate 5 to 8 weeks after embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 and ≤ 36
* Undergoing ovarian stimulation for an In Vitro Fertilization (IVF) or Intra Cytoplasmic Sperm Injection (ICSI)
* Having experienced no more than 1 Embryo Transfer failure
* With basal FSH level ≤ 12 IU/l within the 6 months prior to the study
* Endometrial biopsy during the menstrual cycle preceding the ovarian stimulation (6 to 12 days after a documented ovulation)
* Negative serology for HIV 1 and 2, hepatitis B and C, HTLV 1 and 2, syphilis

Exclusion Criteria:

* Hypersensitivity to one of the culture media components
* Oocyte donation, sperm donation
* Thawed embryos transfer
* Women with endometriosis grade III and IV, chronic endometritis, hydrosalpinx, polycystic ovary, amenorrhoea, anovulation, uterus with malformation, uncontrolled prolactinaemia, uterine synechia, uterine fibroma, women exposed to distilbene, uterine polyps
* Women affected by pathologies associated with any contraindication of being pregnant
* Abnormal gynaecologic bleeding of undetermined origin
* Uncontrolled thyroid (TSH dosage) or adrenal dysfunction
* Neoplasias, any pathologies of the endometrium or the cervix

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 720 (Estimated)
Dates: Start 2008-02

CONTACTS AND LOCATIONS:
Locations (1):
- CMCO, Schiltigheim, France